CLINICAL TRIAL: NCT06905951
Title: The Impact Of Technology In The Myofunctional Therapy Treatment Of Obstructive Sleep Apnea Syndrome
Brief Title: The Impact of Technology in Obstructive Sleep Apnea Myofunctional Therapy
Acronym: OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American Association of Orthodontists Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20231615
Record Dates: First submitted 2025-02-25; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea (OSA); Snoring; Sleep Quality
Keywords: OSA; Myotherapy; Myofunctional Exercises; Snoring; Sleep Apnea; Sleep Quality
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring; Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Both groups receive the same exercise prescription, but one is through a phone application and the other is a piece of paper.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Active Comparator): The mouth exercises are guided and tracked by a phone application.
  Interventions: Other: Exercise
- Analog Group (Active Comparator): The exercise and tracking is done using paper forms.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Mouth, tongue, and throat exercise to strengthen the airway, reducing its collapsibility.
  Other Names: Myofunctional Mouth Exercise

SUMMARY:
This is a study to test if performing airway exercises to improve snoring and sleep apnea using a mobile phone app is better than using a hardcopy guide.

DETAILED DESCRIPTION:
Outcomes will be measured using tone analysis, snoring recording apps, and oximeters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild, moderate, and severe OSA who rejected/failed CPAP or other therapeutic options will be invited to participate in the study.

Exclusion Criteria:

1. Age lower than 18 or higher than 75.
2. BMI > 40
3. Alcoholism or drug abuse
4. A-fib, pacemaker, CHF, strokes, narcotics
5. Neuromuscular disease
6. Use of benzodiazepine hypnotics (may affect muscle tone)
7. Restricted tongue movement
8. Permanently blocked nose
9. TMJ disorder.
10. Lost to follow-up
11. Gained or lost ≥5% of body weight during 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Belun Ring Oxygen Saturation | baseline and then monthly for 3 months.
  Oximeter with pulse rate registration. The oximeter will provide the average level of oxygen saturation in the blood, provided in a percentage outcome.
  .
Belun Ring lowest Oxygen Saturation Level | baseline and then monthly for 3 months.
  Oximeter with pulse rate registration. The oximeter will provide the lowest level of oxygen saturation recorded as a percentage.
Belun Ring Oxygen Saturation under 70% | baseline and then monthly for 3 months.
  Oximeter with pulse rate registration. The oximeter will provide the percentage of sleep that was under 70% SpO2.
Belun Ring AHI | baseline and then monthly for 3 months.
  Oximeter with pulse rate registration. The oximeter provides the Apnea/Hypopnea Index which is the number of apneic events per hour of sleep.
Belun Ring Pulse Rate | baseline and then monthly for 3 months.
  Oximeter with pulse rate registration. The oximeter provides the pulse rate as the average beats per minute with standard deviation, and range.

SECONDARY OUTCOMES:
SnoreLab app | baseline and monthly for 3 months.
  A mobile phone app that records snoring when present, and categorizes into amount and level. Possible outcomes are: none, mild, moderate, severe, and epic.
Tongue Elevation strength | baseline and monthly for 3 months.
  The Iowa Oral Performance Instrument, is a validated intraoral device that measures tongue elevation strength in kPa.
Tongue Protrusion strength | baseline and monthly for 3 months.
  The Iowa Oral Performance Instrument is a validated intraoral device that measures tongue protrusion strength in kPa.
Buccinator strength | baseline and monthly for 3 months.
  The Iowa Oral Performance Instrument is a validated intraoral device that measure the buccinator muscle strength in kPa.
STOP-Bang Questionnaire | baseline and monthly for 3 months.
  STOP-Bang is a validated tool that determines if the subject is at no, low, moderate, or severe risk of sleep-apnea. It provides an objective score that ranges from 0 to 8.
Nasal Obstruction Assessment (NOSE) Questionnaire Score | baseline and monthly for 3 months.
  NOSE is a validated tool that determines the level of difficulty that the subject experienced in breathing through their nose in the past 3 months. The questionnaire provides an objective score stating the risk level that ranges from 0 to 100 with lower scores indicating less nasal blockage and higher scores indicating worse nasal blockage.
PROMIS Sleep Disturbance 8b Short Form Questionnaire | baseline and monthly for 3 months.
  Assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Each question usually has five response options ranging in value from one to five. Values are summed to generate a raw score that is then translated to a t-score with a mean of 50, std of 10.
Epworth Daytime Sleepiness Questionnaire | baseline and monthly for 3 months.
  This is a validated tool that measures a person's daytime sleepiness and is commonly used to help diagnose sleep disorders. Eight prompts with each response scored from 0-3. Higher scores indicates greater sleepiness. It provides an objective score that can range from 0 to 24.
PROMIS Sleep Impairment 8a Short Form Questionnaire | baseline and monthly for 3 months.
  Assesses self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Each question usually has five response options ranging in value from one to five. Values are summed to generate a raw score which is then translated to a t-score with a mean of 50, std of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Palomo, DDS, MSD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University Dental Clinic - Orthodontics, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We intend to publish the results and make them available to the research community. Any additional data is available upon request and will be provided without any PHI.

REFERENCES:
- [Background] Gu W, Leung L, Kwok KC, Wu IC, Folz RJ, Chiang AA. Belun Ring Platform: a novel home sleep apnea testing system for assessment of obstructive sleep apnea. J Clin Sleep Med. 2020 Sep 15;16(9):1611-1617. doi: 10.5664/jcsm.8592. PMID 32464087
- [Background] Baptista PM, Martin F, Ross H, O'Connor Reina C, Plaza G, Casale M. A systematic review of smartphone applications and devices for obstructive sleep apnea. Braz J Otorhinolaryngol. 2022 Nov-Dec;88 Suppl 5(Suppl 5):S188-S197. doi: 10.1016/j.bjorl.2022.01.004. Epub 2022 Feb 4. PMID 35210182
- [Background] Rueda JR, Mugueta-Aguinaga I, Vilaro J, Rueda-Etxebarria M. Myofunctional therapy (oropharyngeal exercises) for obstructive sleep apnoea. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD013449. doi: 10.1002/14651858.CD013449.pub2. PMID 33141943
- [Background] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106
- [Background] Behrents RG, Shelgikar AV, Conley RS, Flores-Mir C, Hans M, Levine M, McNamara JA, Palomo JM, Pliska B, Stockstill JW, Wise J, Murphy S, Nagel NJ, Hittner J. Obstructive sleep apnea and orthodontics: An American Association of Orthodontists White Paper. Am J Orthod Dentofacial Orthop. 2019 Jul;156(1):13-28.e1. doi: 10.1016/j.ajodo.2019.04.009. PMID 31256826
- [Background] Gottlieb DJ, Punjabi NM. Diagnosis and Management of Obstructive Sleep Apnea: A Review. JAMA. 2020 Apr 14;323(14):1389-1400. doi: 10.1001/jama.2020.3514. PMID 32286648

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT06905951/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT06905951/ICF_001.pdf